CLINICAL TRIAL: NCT04864275
Title: Personalized Prediction of Persistent Postsurgical Pain
Acronym: P5
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, simon.haroutounian, Associate Professor, Washington University School of Medicine
Other Study IDs: 202101123
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
P5 is planned as a prospective observational study, collecting evidence-based perioperative data on patient history and demographics, physical function, cognitive measures, psychological, and biological markers associated with increased pain susceptibility, and psychophysical measures of pain processing.

The study will use daily ecologic momentary assessment (EMA) of physical and emotional parameters, and collect data on perioperative events.

Follow up will occur 3 months and 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-75 who are candidates for major surgery (expected surgery duration >1 hour, and expected overnight admission to the hospital), or having one of the following procedures, even if outpatient (total joint replacement, hysterectomy, inguinal hernia repair, breast surgery, or video-assisted thoracic surgery (VATS)).
* Access to a smartphone

Exclusion Criteria:

* Participants who do not speak English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 to 75 years of age and candidates for major surgery at Barnes-Jewish Hospital (expected surgery duration >1h, and expected overnight admission to the hospital, or having one of the following procedures, even if outpatient (total joint replacement, hysterectomy, inguinal hernia repair, breast surgery, or video-assisted thoracic surgery (VATS)) will be approached for consent to this study. Participants will be recruited for participation in the study during their initial preoperative visit to the Center for Perioperative Assessment and Planning (CPAP).
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Persistent Postsurgical Pain (PPSP) | up to 7 months following consent
  Clinically meaningful PPSP will be defined as pain in the surgical area present 3 months after surgery which fulfils one of the following criteria: 1) pain intensity on rest or movement ≥3 on 0-10 numerical rating scale (NRS), or 2) pain interference with any of the seven Brief Pain Inventory items (general activity, mood, walking ability, normal work [including housework], relations with other people, sleep, and enjoyment of life) ≥3 on 0-10 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Associate Professor
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

REFERENCES:
- [Background] Weiser TG, Haynes AB, Molina G, Lipsitz SR, Esquivel MM, Uribe-Leitz T, Fu R, Azad T, Chao TE, Berry WR, Gawande AA. Size and distribution of the global volume of surgery in 2012. Bull World Health Organ. 2016 Mar 1;94(3):201-209F. doi: 10.2471/BLT.15.159293. PMID 26966331
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Derived] Holzer KJ, Alaverdyan H, Xu Z, Frumkin MR, Frey KA, Gregory SH, Rodebaugh TL, Lu C, King CR, Head D, Kannampallil T, Haroutounian S. Protocol for Personalised Prediction of Persistent Postsurgical Pain. BMJ Open. 2026 Feb 4;16(2):e107055. doi: 10.1136/bmjopen-2025-107055. PMID 41638723